CLINICAL TRIAL: NCT00490139
Title: A Randomised, Multi-centre, Open-label, Phase III Study of Adjuvant Lapatinib, Trastuzumab, Their Sequence and Their Combination in Patients With HER2/ErbB2 Positive Primary Breast Cancer
Brief Title: ALTTO (Adjuvant Lapatinib And/Or Trastuzumab Treatment Optimisation) Study; BIG 2-06/N063D
Acronym: ALTTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: North Central Cancer Treatment Group (Network); National Cancer Institute (NCI) (NIH); Breast International Group (Other); Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF106708; CLAP016B2301 (Other: Novartis); 2006-000562-36 (EudraCT Number); NCT00609024 (obsolete NCT alias)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms, Breast
Keywords: Adjuvant; ErbB2-overexpressing; Early stage breast cancer; HER2/neu gene amplified
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lapatinib plus Trastuzumab (Experimental): Design 1: Oral lapatinib 1000 mg daily concurrent with trastuzumab 8 mg/kg IV loading dose followed by 6mg/kg IV every 3 weeks (52 weeks total).
  Design 2: Trastuzumab (4mg/kg loading dose followed by 2mg/kg IV weekly) concurrent with oral lapatinib 750 mg daily and either paclitaxel 80mg/m2 IV weekly for 12 weeks OR docetaxel 75mg/m2 every 21 days for 4 cycles (12 weeks). After completion of chemotherapy, the dose of lapatinib will be increased to 1000mg daily concurrently with trastuzumab every 3 weeks (6mg/kg without loading dose) for an additional 40 weeks (52 weeks total).
  Design 2B: Docetaxel 75mg/m2 and carboplatin AUC 6 every 3 weeks for 6 cycles (18 weeks) administered concurrently with oral lapatinib 750mg plus weekly trastuzumab (4mg/kg IV loading dose followed by 2mg/kg IV. After the completion of chemotherapy, trastuzumab will be administered every 3 weeks (6mg/kg without loading dose) concurrent with lapatinib 1000mg daily for an additional 40 weeks (52 weeks total).
  Interventions: Drug: Lapatinib; Biological: Trastuzumab
- Trastuzumab followed by Lapatinib (Experimental): Design 1: Trastuzumab (4mg/kg IV loading dose followed by 2mg/kg IV weekly) for 12 weeks followed by a 6 week treatment-free interval followed by oral lapatinib 1500mg daily for 34 weeks (52 weeks total).
  Design 2: Trastuzumab (4mg/kg IV loading dose followed by 2mg/kg IV weekly) for 12 weeks administered concomitantly and either paclitaxel 80mg/m2 IV weekly for 12 weeks OR docetaxel 75mg/m2 every 21 days for 4 cycles; followed by a 6 week treatment-free interval followed by oral lapatinib 1500mg daily for 34 weeks (52 weeks total).
  Design 2B: Docetaxel 75mg/m2 and carboplatin AUC 6 every 3 weeks for 6 cycles (18 weeks) administered concomitantly with trastuzumab (4mg/kg IV loading dose followed by 2mg/kg IV weekly) followed by a 6 week treatment-free interval followed by oral lapatinib 1500 mg daily for 28 weeks (52 weeks total).
  Interventions: Drug: Lapatinib; Biological: Trastuzumab
- Lapatinib (Experimental): Design 1: Lapatinib 1500mg oral daily for a total of 52 weeks.
  Design 2: Either paclitaxel 80mg/m2 IV weekly for 12 weeks OR docetaxel 75mg/m2 IV every 3 weeks for 4 cycles administered concomitantly with oral lapatinib at 750mg daily. After completion of chemotherapy, oral lapatinib administered at 1500mg daily for an additional 40 weeks (52 weeks total).
  Design 2B: Docetaxel 75mg/m2 and carboplatin AUC 6 every 3 weeks for 6 cycles (18 weeks) administered concomitantly with oral lapatinib at 750mg daily. After completion of chemotherapy, the dose of lapatinib will be increased to 1500mg oral daily for an additional 40 weeks (52 weeks total).
  Interventions: Drug: Lapatinib
- Trastuzumab (Active Comparator): Design 1: Trastuzumab 8mg/kg IV loading dose followed by 6mg/kg IV every 3 weeks for a total of 52 weeks.
  Design 2: Either paclitaxel 80mg/m2 IV weekly for 12 weeks OR docetaxel 75mg/m2 IV every 3 weeks for 4 cycles administered concomitantly with trastuzumab 4mg/kg IV loading dose followed by 2mg/kg IV weekly. After completion of chemotherapy, trastuzumab administered every 3 weeks (6mg/kg IV without loading dose) for an additional 40 weeks (52 weeks total).
  Design 2B: Docetaxel 75mg/m2 and carboplatin AUC 6 every 3 weeks for 6 cycles (18 weeks) administered concomitantly with trastuzumab 4mg/kg IV loading dose followed by 2mg/kg IV weekly. After completion of chemotherapy, trastuzumab (6mg/kg without loading dose) every 3 weeks for an additional 40 weeks (52 weeks total).
  Interventions: Biological: Trastuzumab

INTERVENTIONS:
Drug: Lapatinib — Small molecule inhibitor
  Other Names: GW572016
  Arms: Lapatinib; Lapatinib plus Trastuzumab; Trastuzumab followed by Lapatinib
Biological: Trastuzumab — Antibody
  Arms: Lapatinib plus Trastuzumab; Trastuzumab; Trastuzumab followed by Lapatinib

SUMMARY:
This was a four-arm (parallel group) randomized, open-label, multicenter Phase 3 study to investigate the use of a combination of Lapatinib and Trastuzumab, a sequence of Trastuzumab followed by Lapatinib, and Lapatinib alone, compared to Trastuzumab alone in the adjuvant treatment of Human Epidermal Growth Factor Receptor 2 (HER2) positive early breast cancer.

DETAILED DESCRIPTION:
Treatment allocation was stratified by blocked randomization, with three stratification factors:

* Hormone receptor status: Estrogen Receptor (ER) and/or Progesterone Receptor (PgR) positive versus both negative.
* Axillary lymph node involvement: not assessed because of neoadjuvant chemotherapy versus node negative versus 1-3 positive nodes versus 4 or more positive nodes.
* Timing of adjuvant chemotherapy: concurrently with taxanes and targeted therapy (Design 2) and concurrently with non-anthracycline-based platinum chemotherapy and targeted therapy (Design 2B) versus all other chemotherapy completed before randomization (Design 1). Treatments delivered differed according to the timing and type of adjuvant chemotherapy.

The primary objective of this study was to compare disease-free survival (DFS) in subjects with HER2 overexpressing and/or amplified breast cancer randomized to trastuzumab for one year versus lapatinib for one year versus trastuzumab (12 or 18 weeks, according to assigned design) followed by a six week treatment-free interval followed by lapatinib (28 or 34 weeks, according to assigned design) versus trastuzumab in combination with lapatinib for one year (52 weeks).

Secondary objectives included treatment comparisons with respect to overall survival, time to recurrence, time to distant recurrence, safety and tolerability, and incidence of brain metastasis.

Based on the recommendation of the Independent Data Monitoring Committee (IDMC) at the first interim analysis (18-Aug-2011), the Lapatinib alone arm was discontinued prior to primary analysis due to futility. The IDMC also stated that the other three arms (trastuzumab alone, sequential trastuzumab/lapatinib arm and the combination arm) could continued as planned with no changes.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients >= 18 years of age with histologically confirmed, non-metastatic, operable and over expression/amplification of HER2 (3+ by IHC and/or FISH positive) primary breast cancer, treated with definitive surgery, with baseline LVEF >= 50%, known hormone receptor status (ER/PgR or ER alone) and ECOG performance status =< 1, were included.
* For Designs 1 and 2: Patients must have had received at least four cycles of an approved anthracycline-based (neo-) adjuvant chemotherapy regimen or a protocol specified exception.
* Approved, signed written informed consent obtained prior to any study specific screening procedures.

Key Exclusion Criteria:

* History of any prior (ipsi- and/or contralateral) invasive breast carcinoma, past (less than 10 years) or current history of malignant neoplasms, any clinically staged T4 tumor, or bilateral tumors.
* Concurrent anti-cancer treatment, except hormonal therapy or radiotherapy for the present breast cancer;
* Patients with positive or suspicious internal mammary nodes identified by sentinel node technique, which had not been irradiated or would not be irradiated, or patients with supraclavicular lymph node involvement.
* Any prior anti-HER therapy, which includes agents that target other members of the HER family of receptors, e.g. gefitinib (Iressa)
* (Neo-) or adjuvant chemotherapy using peripheral stem cell or bone marrow stem cell support;
* Serious cardiac illness or medical conditions.
* Any of the following abnormal laboratory tests immediately prior to randomization:

  1. Serum total bilirubin >1.5 x upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (<2 x ULN) was allowed;
  2. Alanine amino transferase (ALT) or aspartate amino transferase (AST) >2.5 x ULN;
  3. Alkaline phosphatase (ALP) >2.5 x ULN;
  4. Serum creatinine >2.0 x ULN;
  5. Total white blood cell count (WBC) <2.5 x 10^9/L;
  6. Absolute neutrophil count <1.5 x 10^9/L;
  7. Platelets <100 x 10^9/L.
* Women of childbearing potential and male patients with partners of childbearing potential, who are unable or unwilling to use adequate contraceptive measures during study treatment, and pregnant or lactating women.
* Concomitant use of CYP3A4 inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8381 (Actual)
Dates: Start 2007-05-16 (Actual); Primary Completion 2013-12-06 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (766):
- United States (224):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Fairfield, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Martinez, California
  - Novartis Investigative Site, Marysville, California
  - Novartis Investigative Site, Mountain View, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Pleasanton, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Thornton, Colorado
  - Novartis Investigative Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Dover, Delaware
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Lakeland, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Weston, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Columbus, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Lihue, Hawaii
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Evanston, Illinois
  - Novartis Investigative Site, Harvey, Illinois
  - Novartis Investigative Site, Kankakee, Illinois
  - Novartis Investigative Site, Maywood, Illinois
  - Novartis Investigative Site, Mount Vernon, Illinois
  - Novartis Investigative Site, Oak Lawn, Illinois
  - Novartis Investigative Site, Ottawa, Illinois
  - Novartis Investigative Site, Pekin, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Peru, Illinois
  - Novartis Investigative Site, Princeton, Illinois
  - Novartis Investigative Site, Rockford, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Urbana, Illinois
  - Novartis Investigative Site, Beech Grove, Indiana
  - Novartis Investigative Site, Fort Wayne, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Kokomo, Indiana
  - Novartis Investigative Site, Mishawaka, Indiana
  - Novartis Investigative Site, Muncie, Indiana
  - Novartis Investigative Site, South Bend, Indiana
  - Novartis Investigative Site, Ames, Iowa
  - Novartis Investigative Site, Bettendorf, Iowa
  - Novartis Investigative Site, Cedar Rapids, Iowa
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Mason City, Iowa
  - Novartis Investigative Site, Sioux City, Iowa
  - Novartis Investigative Site, Waterloo, Iowa
  - Novartis Investigative Site, Chanute, Kansas
  - Novartis Investigative Site, El Dorado, Kansas
  - Novartis Investigative Site, Independence, Kansas
  - Novartis Investigative Site, Lawrence, Kansas
  - Novartis Investigative Site, Prairie Village, Kansas
  - Novartis Investigative Site, Pratt, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Portland, Maine
  - Novartis Investigative Site, Scarborough, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Bethesda, Maryland
  - Novartis Investigative Site, Frederick, Maryland
  - Novartis Investigative Site, Silver Spring, Maryland
  - Novartis Investigative Site, Towson, Maryland
  - Novartis Investigative Site, Westminster, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Hyannis, Massachusetts
  - Novartis Investigative Site, Peabody, Massachusetts
  - Novartis Investigative Site, Adrian, Michigan
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Dearborn, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Flint, Michigan
  - Novartis Investigative Site, Iron Mountain, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Pontiac, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Saint Joseph, Michigan
  - Novartis Investigative Site, Southfield, Michigan
  - Novartis Investigative Site, Albert Lea, Minnesota
  - Novartis Investigative Site, Duluth, Minnesota
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Mankato, Minnesota
  - Novartis Investigative Site, Maplewood, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Cloud, Minnesota
  - Novartis Investigative Site, Saint Louis Park, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Shakopee, Minnesota
  - Novartis Investigative Site, Waconia, Minnesota
  - Novartis Investigative Site, Willmar, Minnesota
  - Novartis Investigative Site, Pascagoula, Mississippi
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Bozeman, Montana
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Grand Island, Nebraska
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Concord, New Hampshire
  - Novartis Investigative Site, Hooksett, New Hampshire
  - Novartis Investigative Site, Laconia, New Hampshire
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Princeton, New Jersey
  - Novartis Investigative Site, Somerville, New Jersey
  - Novartis Investigative Site, Sparta, New Jersey
  - Novartis Investigative Site, Vineland, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Las Cruces, New Mexico
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Cooperstown, New York
  - Novartis Investigative Site, East Syracuse, New York
  - Novartis Investigative Site, Manhasset, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Hendersonville, North Carolina
  - Novartis Investigative Site, Kinston, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Washington, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Bismarck, North Dakota
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Minot, North Dakota
  - Novartis Investigative Site, Bowling Green, Ohio
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Chillicothe, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Clyde, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Franklin, Ohio
  - Novartis Investigative Site, Greenville, Ohio
  - Novartis Investigative Site, Kettering, Ohio
  - Novartis Investigative Site, Maumee, Ohio
  - Novartis Investigative Site, Sandusky, Ohio
  - Novartis Investigative Site, Sylvania, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Abington, Pennsylvania
  - Novartis Investigative Site, Bethlehem, Pennsylvania
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, Kingston, Pennsylvania
  - Novartis Investigative Site, Nashville, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pottstown, Pennsylvania
  - Novartis Investigative Site, Sayre, Pennsylvania
  - Novartis Investigative Site, West Reading, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Fort Sam Houston, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lackland Air Force Base, Texas
  - Novartis Investigative Site, Longview, Texas
  - Novartis Investigative Site, McAllen, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Midland, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Hampton, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Roanoke, Virginia
  - Novartis Investigative Site, Bellingham, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Charleston, West Virginia
  - Novartis Investigative Site, Huntington, West Virginia
  - Novartis Investigative Site, Appleton, Wisconsin
  - Novartis Investigative Site, Chippewa Falls, Wisconsin
  - Novartis Investigative Site, Eau Claire, Wisconsin
  - Novartis Investigative Site, Green Bay, Wisconsin
  - Novartis Investigative Site, La Crosse, Wisconsin
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Oshkosh, Wisconsin
  - Novartis Investigative Site, Sturgeon Bay, Wisconsin
- Argentina (7):
  - Novartis Investigative Site, Berazategui
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Quilmes
  - Novartis Investigative Site, Rosario
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Australia (32):
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Adelaide
  - Novartis Investigative Site, Bedford Park
  - Novartis Investigative Site, Bunbury
  - Novartis Investigative Site, Campbelltown
  - Novartis Investigative Site, Camperdown
  - Novartis Investigative Site, Coffs Harbour
  - Novartis Investigative Site, Concord
  - Novartis Investigative Site, East Bentleigh
  - Novartis Investigative Site, East Melbourne
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hobart
  - Novartis Investigative Site, Lismore
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Melbourne
  - Novartis Investigative Site, Murdoch
  - Novartis Investigative Site, Nambour
  - Novartis Investigative Site, Nedlands
  - Novartis Investigative Site, North Sydney
  - Novartis Investigative Site, Parkville
  - Novartis Investigative Site, Port Macquarie
  - Novartis Investigative Site, Randwick
  - Novartis Investigative Site, South Brisbane
  - Novartis Investigative Site, Subiaco
  - Novartis Investigative Site, Taree
  - Novartis Investigative Site, Tweed Heads
  - Novartis Investigative Site, Wagga Wagga
  - Novartis Investigative Site, Waratah
  - Novartis Investigative Site, Wendouree
  - Novartis Investigative Site, Westmead
  - Novartis Investigative Site, Woodville
  - Novartis Investigative Site, Woolloongabba
- Austria (5):
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Steyr
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Villach
- Belgium (25):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Haine-Saint-Paul
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Mons
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Sint-Niklaas
  - Novartis Investigative Site, Tournai
  - Novartis Investigative Site, Turnhout
  - Novartis Investigative Site, Verviers
  - Novartis Investigative Site, Wilrijk
  - Novartis Investigative Site, Yvoir
- Brazil (7):
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, Belo Horizonte
  - Novartis Investigative Site, Porte Alegre
  - Novartis Investigative Site, Porto Alegre
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Salvador
  - Novartis Investigative Site, Santo André
- Bulgaria (3):
  - Novartis Investigative Site, Shumen
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (10):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Charlottetown
  - Novartis Investigative Site, Kelowna
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Moncton
  - Novartis Investigative Site, Regina
  - Novartis Investigative Site, Sault Ste. Marie
  - Novartis Investigative Site, Sherbrooke
  - Novartis Investigative Site, St. Catharines
  - Novartis Investigative Site, Vancouver
- Chile (5):
  - Novartis Investigative Site, Santiago
  - Novartis Investigative Site, Temuco
  - Novartis Investigative Site, Valdivia
  - Novartis Investigative Site, Valparaíso
  - Novartis Investigative Site, Viña del Mar
- China (4):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Czechia (8):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Chomutov
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Ústí nad Labem
- Denmark (11):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Arhus C
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Hilleroed
  - Novartis Investigative Site, Koebenhavn Oe
  - Novartis Investigative Site, Næstved
  - Novartis Investigative Site, Odense
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Vejle
  - Novartis Investigative Site, Viborg
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (42):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Annecy
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Béthune
  - Novartis Investigative Site, Brive-la-Gaillarde
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Coudekerque-Branche
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Draguignan
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Hyères
  - Novartis Investigative Site, La Seyne-sur-Mer
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Mont-de-Marsan
  - Novartis Investigative Site, Montbéliard
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perin Sur Mer
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Périgueux
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Cloud
  - Novartis Investigative Site, Saint-Grégoire
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Saint-Jean
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Valenciennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (135):
  - Novartis Investigative Site, Ansbach
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Aschersleben
  - Novartis Investigative Site, Aurich
  - Novartis Investigative Site, Bad Oldesloe
  - Novartis Investigative Site, Bad Reichenhall
  - Novartis Investigative Site, Baden-Baden
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Bergisch Gladbach
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Brandenburg
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cuxhaven
  - Novartis Investigative Site, Dachau
  - Novartis Investigative Site, Deggendorf
  - Novartis Investigative Site, Donauwörth
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eggenfelden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Eschweiler
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Flensburg
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Garmisch-Partenkirchen
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göppingen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Güstrow
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamelin
  - Novartis Investigative Site, Hamm-Heessen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heide
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Hoyerswerda
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kempten
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Konstanz
  - Novartis Investigative Site, Landshut
  - Novartis Investigative Site, Landstuhl
  - Novartis Investigative Site, Leer
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Limburg
  - Novartis Investigative Site, Loerrach
  - Novartis Investigative Site, Luckenwalde
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Ludwigsfelde
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marktredwitz
  - Novartis Investigative Site, Meiningen
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Mutlangen
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Olpe
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Ostfildern
  - Novartis Investigative Site, Porta Westfalica
  - Novartis Investigative Site, Radebeul
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Rendsburg
  - Novartis Investigative Site, Reutlingen
  - Novartis Investigative Site, Rheinfelden
  - Novartis Investigative Site, Rodewisch
  - Novartis Investigative Site, Rosenheim
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rotenburg (Wümme)
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schkeuditz
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Sigmaringen
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stadthagen
  - Novartis Investigative Site, Stendal
  - Novartis Investigative Site, Stralsund
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Torgau
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Vechta
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Villingen-Schwenningen
  - Novartis Investigative Site, Weißenfels
  - Novartis Investigative Site, Wesel
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würselen
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zittau
  - Novartis Investigative Site, Zwickau
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Hong Kong (2):
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Tuenmen
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Szeged
- India (7):
  - Novartis Investigative Site, Gūrgaon
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, Kolkata
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, Nagpur
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Trivandrum
- Ireland (3):
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
- Israel (8):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Netanya
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Zrifin
- Italy (40):
  - Novartis Investigative Site, Asti
  - Novartis Investigative Site, Avellino
  - Novartis Investigative Site, Aviano
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Biella
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Brindisi
  - Novartis Investigative Site, Candiolo
  - Novartis Investigative Site, Carpi
  - Novartis Investigative Site, Cosenza
  - Novartis Investigative Site, Cremona
  - Novartis Investigative Site, Fano
  - Novartis Investigative Site, Fermo
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Lecce
  - Novartis Investigative Site, Lecco
  - Novartis Investigative Site, Lido di Camaiore
  - Novartis Investigative Site, Livorno
  - Novartis Investigative Site, Mantova
  - Novartis Investigative Site, Meldola
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Monserrato
  - Novartis Investigative Site, Monza
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Poggibonsi
  - Novartis Investigative Site, Potenza
  - Novartis Investigative Site, Prato
  - Novartis Investigative Site, Ragusa
  - Novartis Investigative Site, Ravenna
  - Novartis Investigative Site, Rimini
  - Novartis Investigative Site, Rozzano
  - Novartis Investigative Site, San Fermo della Battaglia
  - Novartis Investigative Site, Saronno
  - Novartis Investigative Site, Sassari
  - Novartis Investigative Site, Trento
  - Novartis Investigative Site, Treviglio
  - Novartis Investigative Site, Udine
  - Novartis Investigative Site, Varese
  - Novartis Investigative Site, Viterbo
- Japan (10):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Ibaraki
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Tokyo
- Mexico (4):
  - Novartis Investigative Site, Chihuahua City
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, México
  - Novartis Investigative Site, Toluca
- Netherlands (16):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Hilversum
  - Novartis Investigative Site, Hoogeveen
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Leidschendam
  - Novartis Investigative Site, Purmerend
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Tilburg
  - Novartis Investigative Site, Utrecht
- New Zealand (3):
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Palmerston North
  - Novartis Investigative Site, Wellington
- Norway (2):
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Tromsø
- Pakistan (3):
  - Novartis Investigative Site, Karachi
  - Novartis Investigative Site, Lahore
  - Novartis Investigative Site, Rawalpindi
- Peru (2):
  - Novartis Investigative Site, Callao
  - Novartis Investigative Site, Lima
- Philippines (4):
  - Novartis Investigative Site, Cebu
  - Novartis Investigative Site, Quezon City
  - Novartis Investigative Site, Sampaloc
  - Novartis Investigative Site, San Juan City
- Poland (10):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Romania (3):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Iași
- Russia (13):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Voronezh
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (4):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Žilina
- Novartis Investigative Site, Ljubljana, Slovenia
- South Africa (7):
  - Novartis Investigative Site, Capital Park
  - Novartis Investigative Site, Groenkloof
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Observatory
  - Novartis Investigative Site, Panorama
  - Novartis Investigative Site, Parktown
  - Novartis Investigative Site, Pretoria
- South Korea (3):
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (29):
  - Novartis Investigative Site, Alcoy
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Cadiz
  - Novartis Investigative Site, Castellon
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Elda
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Lugo
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Mataró
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Móstoles
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Santa Cruz de Tenerife
  - Novartis Investigative Site, Santander
  - Novartis Investigative Site, Santiago
  - Novartis Investigative Site, Segovia
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Tarrasa, Barcelona
  - Novartis Investigative Site, Toledo
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Vizcaya
  - Novartis Investigative Site, Zamora
- Switzerland (9):
  - Novartis Investigative Site, Aarau
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bellinzona
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Locarno
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Thun
  - Novartis Investigative Site, Zurich
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan County
  - Novartis Investigative Site, Taipei
- Thailand (5):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Phitsanulok
  - Novartis Investigative Site, Songkhla
- Ukraine (7):
  - Novartis Investigative Site, Chernivtsi
  - Novartis Investigative Site, Donetsk
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Simferopol
  - Novartis Investigative Site, Uzhhorod
- United Kingdom (39):
  - Novartis Investigative Site, Canterbury, Kent
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Brighton
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chelmsford
  - Novartis Investigative Site, Cheltenham
  - Novartis Investigative Site, Cottingham
  - Novartis Investigative Site, Dorchester
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Grimsby
  - Novartis Investigative Site, Guildford
  - Novartis Investigative Site, Gwynedd
  - Novartis Investigative Site, Huddersfield
  - Novartis Investigative Site, Ipswich
  - Novartis Investigative Site, Lancaster
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Maidstone
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Northwood
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Prittlewell Chase
  - Novartis Investigative Site, Romford
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Shrewsbury
  - Novartis Investigative Site, St Helens
  - Novartis Investigative Site, Stoke-on-Trent
  - Novartis Investigative Site, Sutton
  - Novartis Investigative Site, Swansea
  - Novartis Investigative Site, Worthing

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rediti M, Venet D, Joaquin Garcia A, Maetens M, Vincent D, Majjaj S, El-Abed S, Di Cosimo S, Ueno T, Izquierdo M, Piccart M, Pusztai L, Loi S, Salgado R, Viale G, Rothe F, Sotiriou C. Identification of HER2-positive breast cancer molecular subtypes with potential clinical implications in the ALTTO clinical trial. Nat Commun. 2024 Nov 29;15(1):10402. doi: 10.1038/s41467-024-54621-3. PMID 39613746
- [Derived] Nader-Marta G, Debien V, Eiger D, Tsourti Z, Caparica R, Kassapian M, Napoleone S, Hultsch S, Korde L, Wang Y, Chumsri S, Pritchard KI, Untch M, Bellet-Ezquerra M, Dornelles Rosa D, Moreno-Aspitia A, Piccart M, Dafni U, de Azambuja E. Outcomes of patients with small and node-negative HER2-positive early breast cancer treated with adjuvant chemotherapy and anti-HER2 therapy-a sub-analysis of the ALTTO study. Br J Cancer. 2022 Nov;127(10):1799-1807. doi: 10.1038/s41416-022-01963-8. Epub 2022 Sep 1. PMID 36050448
- [Derived] Moreno-Aspitia A, Holmes EM, Jackisch C, de Azambuja E, Boyle F, Hillman DW, Korde L, Fumagalli D, Izquierdo MA, McCullough AE, Wolff AC, Pritchard KI, Untch M, Guillaume S, Ewer MS, Shao Z, Sim SH, Aziz Z, Demetriou G, Mehta AO, Andersson M, Toi M, Lang I, Xu B, Smith IE, Barrios CH, Baselga J, Gelber RD, Piccart-Gebhart M; ALTTO Steering Committee and Investigators. Updated results from the international phase III ALTTO trial (BIG 2-06/Alliance N063D). Eur J Cancer. 2021 May;148:287-296. doi: 10.1016/j.ejca.2021.01.053. Epub 2021 Mar 23. PMID 33765513
- [Derived] Sonnenblick A, Agbor-Tarh D, de Azambuja E, Hultsch S, Izquierdo M, Liu M, Pruneri G, Harbeck N, Piccart M, Moreno-Aspita A, Granit RZ, Rouas G, Fahoum I, Sotiriou C. STAT3 activation in HER2-positive breast cancers: Analysis of data from a large prospective trial. Int J Cancer. 2021 Mar 15;148(6):1529-1535. doi: 10.1002/ijc.33385. Epub 2020 Nov 23. PMID 33152119
- [Derived] Eiger D, Ponde NF, Agbor-Tarh D, Moreno-Aspitia A, Piccart M, Hilbers FS, Werner O, Chumsri S, Dueck A, Kroep JR, Gomez H, Lang I, Rodeheffer RJ, Ewer MS, Suter T, de Azambuja E. Long-term cardiac outcomes of patients with HER2-positive breast cancer treated in the adjuvant lapatinib and/or trastuzumab Treatment Optimization Trial. Br J Cancer. 2020 May;122(10):1453-1460. doi: 10.1038/s41416-020-0786-x. Epub 2020 Mar 16. PMID 32203207
- [Derived] Holmes EM, Bradbury I, Williams LS, Korde L, de Azambuja E, Fumagalli D, Moreno-Aspitia A, Baselga J, Piccart-Gebhart M, Dueck AC, Gelber RD; ALTTO Trial Study Team. Are we assuming too much with our statistical assumptions? Lessons learned from the ALTTO trial. Ann Oncol. 2019 Sep 1;30(9):1507-1513. doi: 10.1093/annonc/mdz195. PMID 31240310
- [Derived] McCullough AE, Dell'orto P, Reinholz MM, Gelber RD, Dueck AC, Russo L, Jenkins RB, Andrighetto S, Chen B, Jackisch C, Untch M, Perez EA, Piccart-Gebhart MJ, Viale G. Central pathology laboratory review of HER2 and ER in early breast cancer: an ALTTO trial [BIG 2-06/NCCTG N063D (Alliance)] ring study. Breast Cancer Res Treat. 2014 Feb;143(3):485-92. doi: 10.1007/s10549-013-2827-0. Epub 2014 Jan 7. PMID 24395109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 969 centers in 44 countries worldwide.
Pre-assignment Details: Based on the IDMC results from 18 August 2011, any patient enrolled onto Lapatinib arm were considered for a new treatment strategy based on discussion with their physician.
Groups:
- Lapatinib Plus Trastuzumab: Participants received treatment per one of three designs and adjuvant radiotherapy / adjuvant anti-estrogen therapy when clinically indicated.
  * Design 1: oral lapatinib (OL) 1000 milligrams (mg) daily with trastuzumab (tras) (8 milligrams per kilogram [mg/kg] intravenous [IV] loading dose [LD], followed by 6 mg/kg IV every 3 weeks [E3W]) for 52 weeks (wks).
  * Design 2: OL 750 mg daily plus wkly tras (4 mg/kg LD, followed by 2 mg/kg IV) concomitantly (conc.) with wkly paclitaxel (pac) 80 mg per squared meter (mg/m^2) IV or docetaxel (doc) 75 mg/m^2 IV E3W for 12 wks. After completion of pac or doc, par. received OL at an increased dose of 1000 mg daily in combination with tras (6 mg/kg without a LD) E3W for 40 wks.
  * Design 2B: OL 750 mg plus wkly tras (4 mg/kg IV LD, followed by 2 mg/kg IV wkly) conc. with doc 75 mg/m^2 E3W and carboplatin (carb) AUC6 IV for 18 wks. After completion of doc and carb, par. received tras E3W (6 mg/kg without a LD) plus OL 1000 mg daily for 34 wks.
- Trastuzumab Followed by Lapatinib: Participants received treatment per one of three designs and adjuvant radiotherapy / adjuvant anti-estrogen therapy when clinically indicated.
  * Design 1: weekly tras for 12 weeks (4 mg/kg IV loading dose, followed by 2 mg/kg IV weekly), followed by a 6-week washout period, followed by oral lap 1500 mg daily for 34 weeks.
  * Design 2: weekly tras (4 mg/kg IV loading dose, followed by 2 mg/kg IV) concomitantly with weekly paclitaxel 80 mg/m^2 IV or docetaxel 75 mg/m^2 IV every 3 weeks for 12 weeks, followed by a 6-week washout period, followed by oral lap 1500 mg daily for 34 weeks.
  * Design 2B: weekly tras (4 mg/kg IV loading dose, followed by 2 mg/kg IV weekly) concomitantly with docetaxel 75 mg/m^2 every 3 weeks and carboplatin AUC6 IV for 18 weeks, followed by a 6-week washout period, followed by oral lap 1500 mg daily for 28 weeks.
- Lapatinib: Participants received treatment per one of three designs and adjuvant radiotherapy / adjuvant anti-estrogen therapy when clinically indicated.
  * Design 1: oral lap 1500 mg daily for 52 weeks.
  * Design 2: oral lap 750 mg daily concomitantly with weekly paclitaxel 80 mg/m^2 IV or docetaxel 75 mg/m^2 IV every 3 weeks, for 12 weeks. After completion of paclitaxel or docetaxel, participants received oral lap at an increased dose of 1500 mg daily for 40 weeks.
  * Design 2B: oral lap 750 mg daily concomitantly with docetaxel 75 mg/m^2 every 3 weeks and carboplatin AUC6 IV, for 18 weeks. After completion of docetaxel and carboplatin, oral lap was given at an increased dose of 1500 mg for 34 weeks.
- Trastuzumab: Participants received treatment per one of three designs and adjuvant radiotherapy / adjuvant anti-estrogen therapy when clinically indicated.
  * Design 1: tras 8 mg/kg IV LD, followed by 6 mg/kg IV every 3 weeks for 52 weeks.
  * Design 2: weekly tras (4 mg/kg IV LD, followed by 2 mg/kg IV weekly) concomitantly with weekly paclitaxel 80 mg/m^2 IV or docetaxel 75 mg/m^2 IV every 3 weeks, for 12 weeks. After completion of paclitaxel or docetaxel, participants received tras (6 mg/kg without a LD every 3 weeks for 40 weeks.
  * Design 2B: weekly tras (4 mg/kg IV LD, followed by 2 mg/kg IV weekly) concomitantly with docetaxel 75 mg/m^2 every 3 weeks and carboplatin AUC6 IV, for 18 weeks. After completion of docetaxel and carboplatin, participants received tras every 3 weeks (6 mg/kg without a LD) for 34 weeks. "
Period: Overall Study
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Started (All randomized participants were included in the Intent-to-Treat (IIT) Population) | 2093 | 2091 | 2100 | 2097
Safety Population (All randomized participants who were administered at least one dose of investigational targeted treatment) | 2061 | 2076 | 2056 | 2076
Completed (Deaths and participants who completed survival follow-up) | 1132 | 1184 | 1179 | 1192
Not Completed | 961 | 907 | 921 | 905
Not completed — Lost to Follow-up | 249 | 216 | 205 | 229
Not completed — Withdrawal by Subject | 333 | 322 | 396 | 295
Not completed — Patient did not sign ICF 12 | 169 | 176 | 139 | 167
Not completed — Data unavailable due to regulatory issues | 98 | 96 | 85 | 95
Not completed — Data unavailable due to lapsed ethical consent | 14 | 13 | 14 | 14
Not completed — Other reasons as defined per protocol | 98 | 84 | 82 | 105

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab | Total
Number analyzed (Participants) | 2093 | 2091 | 2100 | 2097 | 8381
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (10.23) | 50.8 (10.32) | 51.2 (10.18) | 51.0 (10.25) | 51.0 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2091 | 2086 | 2098 | 2097 | 8372
  Male | 2 | 5 | 2 | 0 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 48 | 45 | 47 | 47 | 187
  Asian: Central/South | 107 | 103 | 110 | 109 | 429
  Asian: East | 311 | 312 | 299 | 314 | 1236
  Asian: Japanese | 33 | 36 | 33 | 43 | 145
  Asian: South East | 95 | 92 | 107 | 89 | 383
  Black or African American | 38 | 30 | 43 | 25 | 136
  Native Hawaiian or Other Pacific | 2 | 4 | 4 | 5 | 15
  White: Arabic | 53 | 52 | 62 | 69 | 236
  White: Caucasian | 1392 | 1402 | 1372 | 1382 | 5548
  Other Race | 14 | 14 | 23 | 14 | 65
  Unknown/Missing | 0 | 1 | 0 | 0 | 1
Hormone Receptor (HR) Status [Count of Participants; unit: Participants] — HR status was determined from the percentage of Estrogen Receptor (ER) and Progesterone Receptor (PgR) cells stained positive: a) Positive: if the percentage of cells stained positive is >= 1% for either ER or PgR; b) Negative: if the percentage of cells stained positive is < 1% for both ER and PgR
  Participants
    Negative | 890 | 886 | 903 | 897 | 3576
    Positive | 1203 | 1205 | 1197 | 1200 | 4805
Timing of Chemotherapy [Count of Participants; unit: Participants] — Timing of (neo)adjuvant chemotherapy was defined as follows: Design 1 - sequentially (all chemotherapy completed prior to randomization) versus Design 2 - concurrently with targeted therapy (taxane medication administered with targeted treatment after randomization). Subjects treated concurrently but without anthracycline (Design 2B) were regarded as part of Design 2 for all stratified analyses.
  Participants
    Sequential | 1155 | 1143 | 1168 | 1147 | 4613
    Concurrent | 938 | 948 | 932 | 950 | 3768
Axillary Lymph Node Status [Count of Participants; unit: Participants] — Axillary Lymph Node Status was categorized as: a) Not applicable (neoadjuvant chemotherapy); b) Node negative (no neoadjuvant chemotherapy); c) 1-3 positive nodes (no neoadjuvant chemotherapy); d) >= 4 positive nodes (no neoadjuvant chemotherapy)
  Participants
    Not applicable (neoadjuvant chemotherapy) | 168 | 170 | 167 | 181 | 686
    Node negative (no neoadjuvant chemotherapy) | 845 | 842 | 841 | 844 | 3372
    1-3 positive nodes (no neoadjuvant chemotherapy) | 617 | 617 | 620 | 603 | 2457
    >= 4 positive nodes (no neoadjuvant chemotherapy) | 463 | 462 | 472 | 469 | 1866

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS) at the Primary Analysis
Description: Disease-Free Survival (DFS) was defined as the interval between randomization and the date of first occurrence of disease recurrence (local, regional or distant), a contralateral invasive breast cancer, a second primary cancer or death without recurrence. Only deaths occurring in participants whose clinical follow-up was ongoing at the time of death and who had no recurrence, contralateral breast cancer (CBC) or second primary malignancy (SPM) reported prior to death were considered as death without recurrence. DFS was estimated using the Kaplan Meier method. The percentile data values presented here indicate the percentage (95, 90, 85, 80 and 75 percent) of participants who had disease free survival for the indicated years.
Time Frame: From randomization until the date of the first occurrence of disease recurrence, a contralateral invasive breast cancer, a second primary cancer, or death from any cause (median follow-up of 4.5 years)
Population: Intent-to-Treat (ITT) Population. DFS data for the Lapatinib alone arm include date collected up to the first interim analysis (data cut-off 11th July 2011), as the Lapatinib arm was discontinued prior to the primary analysis due to futility. All the other arms include data up to median follow-up of 4.5 years.
Measure: Number; unit: Years
Groups:
- Lapatinib: Participants received treatment per one of the following three designs. Design 1: oral lap 1500 mg daily for 52 weeks. Design 2: oral lap 750 mg daily concomitantly with weekly paclitaxel 80 mg/m^2 IV or docetaxel 75 mg/m^2 IV every 3 weeks, for 12 weeks. After completion of paclitaxel or docetaxel, participants received oral lap at an increased dose of 1500 mg daily for 40 weeks. Design 2B: oral lap 750 mg daily concomitantly with docetaxel 75 mg/m^2 every 3 weeks and carboplatin AUC6 IV, for 18 weeks. After completion of docetaxel and carboplatin, oral lap was given at an increased dose of 1500 mg for 34 weeks. Participants also received adjuvant radiotherapy and adjuvant anti-estrogen therapy when clinically indicated.
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 2100 | 2097
Years
  95th Percentile | 1.9 | 1.3 | 1.0 | 1.5
  90th Percentile | 3.2 | 2.8 | 1.8 | 2.6
  85th Percentile | 5.1 | 4.8 | 2.8 | 4.2
  80th Percentile | 6.1 | NA — There were not enough data (insufficient follow-up) to be able to compute this data point. | NA — DFS data for the Lapatinib alone arm include date collected up to the first interim analysis (data cut-off 11th July 2011), as the Lapatinib arm was discontinued prior to the primary analysis due to futility | 5.6
  75th Percentile | 6.1 | NA — There were not enough data (insufficient follow-up) to be able to compute this data point. | NA — DFS data for the Lapatinib alone arm include date collected up to the first interim analysis (data cut-off 11th July 2011), as the Lapatinib arm was discontinued prior to the primary analysis due to futility | NA — There were not enough data (insufficient follow-up) to be able to compute this data point.
Statistical Analysis 1: Comparison: Lapatinib Plus Trastuzumab vs Trastuzumab; Test type: Superiority or Other; p = 0.048, Log Rank; Stratification was by chemotherapy timing, hormone receptor status, and axillary lymph node status; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 1.00] — The estimate of the treatment hazard ratio (lap plus tras versus tras) was based on the Cox proportional hazards model adjusting for the stratification factors of chemotherapy timing, hormone receptor status, and axillary lymph node status
Statistical Analysis 2: Comparison: Trastuzumab Followed by Lapatinib vs Trastuzumab; Test type: Superiority or Other; p = 0.610, Log Rank; Stratification was by chemotherapy timing, hormone receptor status, and axillary lymph node status; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.81 to 1.13] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Disease-Free Survival (DFS) at the 10-Year Follow-Up
Description: Disease-Free Survival (DFS) was defined as the interval between randomization and the date of first occurrence of disease recurrence (local, regional or distant), a contralateral invasive breast cancer, a second primary cancer or death without recurrence. Only deaths occurring in participants whose clinical follow-up was ongoing at the time of death and who had no recurrence, contralateral breast cancer (CBC) or second primary malignancy (SPM) reported prior to death were considered as death without recurrence. DFS was estimated using the Kaplan Meier method. The percentile data values presented here indicate the percentage (95, 90, 85 and 80 percent) of participants who had disease free survival for the indicated years.
Time Frame: From randomization until the date of the first occurrence of disease recurrence, a contralateral invasive breast cancer, a second primary cancer, or death from any cause, assessed up to approximately 10 years
Population: Intent-to-Treat (ITT) Population. The Lapatinib alone arm was discontinued prior to primary analysis due to futility.
Measure: Number; unit: Years
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 0 | 2097
Years
  95th Percentile | 1.89 | 1.27 |  | 1.49
  90th Percentile | 3.21 | 2.80 |  | 2.63
  85th Percentile | 5.92 | 4.85 |  | 4.43
  80th Percentile | 8.99 | 9.18 |  | 7.42
Statistical Analysis 1: Comparison: Lapatinib Plus Trastuzumab vs Trastuzumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.887, 95% CI 2-sided [0.77 to 1.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Trastuzumab Followed by Lapatinib vs Trastuzumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.914, 95% CI 2-sided [0.80 to 1.05] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival (OS) at the Primary Analysis
Description: Overall Survival (OS) was defined as the time from randomization until death due to any cause. Participants who had not died were censored at the last date they were known to be alive, or date of withdrawal of consent. OS was calculated in years as (date of death minus the date of randomization +1) divided by 365.25. The percentile data values presented here indicate the percentage (99, 98, 97, 96, 95 and 90 percent) of participants who survived for the indicated years.
Time Frame: From randomization until death due to any cause (median follow-up of 4.5 years)
Population: Intent-to-Treat (ITT) Population. Zero participants were analyzed in the lapatinib arm, as the Independent Data Monitoring Committee discontinued the lapatinib-alone arm due to futility at the time of the first interim analysis (lapatinib participants were then offered trastuzumab).
Measure: Number; unit: Years
Groups:
- Lapatinib: Participants received treatment per one of the following three designs. Design 1: oral lap 1500 mg daily for 52 weeks.
  Design 2: oral lap 750 mg daily concomitantly with weekly paclitaxel 80 mg/m^2 IV or docetaxel 75 mg/m^2 IV every 3 weeks, for 12 weeks. After completion of paclitaxel or docetaxel, participants received oral lap at an increased dose of 1500 mg daily for 40 weeks. Design 2B: oral lap 750 mg daily concomitantly with docetaxel 75 mg/m^2 every 3 weeks and carboplatin AUC6 IV, for 18 weeks. After completion of docetaxel and carboplatin, oral lap was given at an increased dose of 1500 mg for 34 weeks. Participants also received adjuvant radiotherapy and adjuvant antiestrogen therapy when clinically indicated.
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 0 | 2097
Years
  99th Percentile | 1.7 | 1.2 |  | 1.7
  98th Percentile | 2.2 | 1.6 |  | 2.1
  97th Percentile | 2.8 | 2.2 |  | 2.6
  96th Percentile | 3.4 | 2.9 |  | 3.0
  95th Percentile | 3.9 | 3.7 |  | 3.6
  90th Percentile | NA — There were not enough data (insufficient follow-up) to be able to compute this data point. | NA — There were not enough data (insufficient follow-up) to be able to compute this data point. |  | 5.9
Statistical Analysis 1: Comparison: Lapatinib Plus Trastuzumab vs Trastuzumab; Test type: Superiority or Other; p = 0.078, Log Rank; Stratification was by chemotherapy timing, hormone receptor status, and axillary lymph node status; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.62 to 1.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Trastuzumab Followed by Lapatinib vs Trastuzumab; Test type: Superiority or Other; p = 0.433, Log Rank; Stratification was by chemotherapy timing, hormone receptor status, and axillary lymph node status; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.71 to 1.16] — The estimate of the treatment hazard ratio (tras followed by lap versus tras) was based on the Cox proportional hazards model adjusting for the stratification factors of chemotherapy timing, hormone receptor status, and axillary lymph node status

4. Secondary Outcome: Overall Survival (OS) at the 10-Year Follow-Up
Description: Overall Survival (OS) was defined as the time from randomization until death due to any cause. Participants who had not died were censored at the last date they were known to be alive, or date of withdrawal of consent. OS was calculated in years as (date of death minus the date of randomization +1) divided by 365.25. The percentile data values presented here indicate the percentage (99, 98, 95 and 90 percent) of participants who survived for the indicated years.
Time Frame: From randomization until death due to any cause, assessed up to approximately 10 years
Population: Intent-to-Treat (ITT) Population. The Lapatinib alone arm was discontinued prior to primary analysis due to futility.
Measure: Number; unit: Years
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 0 | 2097
Years
  99th Percentile | 1.68 | 1.17 |  | 1.75
  98th Percentile | 2.19 | 1.60 |  | 2.07
  95th Percentile | 3.92 | 3.52 |  | 3.65
  90th Percentile | 8.31 | 8.49 |  | 6.72
Statistical Analysis 1: Comparison: Lapatinib Plus Trastuzumab vs Trastuzumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.853, 95% CI 2-sided [0.70 to 1.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Trastuzumab Followed by Lapatinib vs Trastuzumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.863, 95% CI 2-sided [0.71 to 1.04] — [estimate comment as in outcome 3, analysis 2]

5. Secondary Outcome: Analysis of Time to Recurrence (TTR)
Description: Time to Recurrence (TTR) was defined as the the time from randomization to breast cancer recurrence, ignoring second primary cancers (including contralateral breast cancers and non-breast second malignancies) and counting deaths without recurrence as a competing risk.
Time Frame: From randomization until the date of the first occurrence of a disease recurrence, assessed up to approximately 10 years
Population: Intent-to-Treat (ITT) Population. The Lapatinib alone arm was discontinued prior to primary analysis due to futility.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 0 | 2097
Participants
  Local, regional, or distant recurrence | 243 | 275 |  | 298
  Death as a competing risk | 43 | 38 |  | 46
  Censored | 1807 | 1778 |  | 1753
Statistical Analysis 1: Comparison: Lapatinib Plus Trastuzumab vs Trastuzumab; Test type: Superiority or Other — Time to recurrence was analyzed using competing risks methodology with death (without event) as a competing risk; Hazard Ratio (HR) = 0.811, 95% CI 2-sided [0.68 to 0.96]
Statistical Analysis 2: Comparison: Trastuzumab Followed by Lapatinib vs Trastuzumab; Test type: Superiority or Other — Time to recurrence was analyzed using competing risks methodology with death (without event) as a competing risk; Hazard Ratio (HR) = 0.930, 95% CI 2-sided [0.79 to 1.10]

6. Secondary Outcome: Analysis of Time to Distant Recurrence (TTDR)
Description: Time to Distant Recurrence (TTDR) was defined as the the time from randomization to first distant breast cancer recurrence, ignoring locoregional recurrences and second primary cancers, (including contralateral breast cancers and non-breast second malignancies ) and counting deaths without recurrence as a competing risk.
Time Frame: From randomization until the date of the first occurrence of distant recurrence, assessed up to approximately 10 years
Population: Intent-to-Treat (ITT) Population. The Lapatinib alone arm was discontinued prior to primary analysis due to futility.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 0 | 2097
Participants
  Distant recurrence | 213 | 238 |  | 250
  Death as a competing risk | 45 | 41 |  | 54
  Censored | 1835 | 1812 |  | 1793
Statistical Analysis 1: Comparison: Lapatinib Plus Trastuzumab vs Trastuzumab; Test type: Superiority or Other — Time to distant recurrence was analyzed using competing risks methodology with death (without event) as a competing risk; Hazard Ratio (HR) = 0.852, 95% CI 2-sided [0.71 to 1.02]
Statistical Analysis 2: Comparison: Trastuzumab Followed by Lapatinib vs Trastuzumab; Test type: Superiority or Other — [test comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.81 to 1.16]

7. Secondary Outcome: Analysis of Time to Central Nervous System (CNS) Recurrence
Description: Time to Central Nervous System (CNS) recurrence was defined as the time from randomization to first CNS recurrence. Both brain metastasis and meningitis carcinomatosa were considered.
Time Frame: From randomization until the first central nervous system recurrence, assessed up to approximately 10 years
Population: Intent-to-Treat (ITT) Population. The Lapatinib alone arm was discontinued prior to primary analysis due to futility.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 0 | 2097
Participants
  CNS recurrence | 91 | 91 |  | 95
  Death as a competing risk | 114 | 117 |  | 142
  Censored | 1888 | 1883 |  | 1860
Statistical Analysis 1: Comparison: Lapatinib Plus Trastuzumab vs Trastuzumab; Test type: Superiority or Other — Time to CNS recurrence was analyzed using competing risks methodology with death (without event) as a competing risk; Hazard Ratio (HR) = 0.986, 95% CI 2-sided [0.74 to 1.31]
Statistical Analysis 2: Comparison: Trastuzumab Followed by Lapatinib vs Trastuzumab; Test type: Superiority or Other — Time to CNS recurrence was analyzed using competing risks methodology with death (without event) as a competing risk; Hazard Ratio (HR) = 0.980, 95% CI 2-sided [0.74 to 1.31]

8. Secondary Outcome: Cumulative Incidence of Brain Metastases
Description: The cumulative incidence of brain metastases as the first site of breast cancer recurrence among treatment arms was assessed using a hierarchy of primary type and location of first DFS event in cases where more than one event was identified simultaneously. Because diagnostic procedures for different types of recurrence could not be performed on exactly the same day, any diagnoses noted within a two month (60 day) period of the first reported event was considered as identified simultaneously for purposes of defining the type of the first event and the date of event was be regarded as the earliest of the relevant events.
Time Frame: as for outcome 5
Population: Intent-to-Treat (ITT) Population. The Lapatinib alone arm was discontinued prior to primary analysis due to futility.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 0 | 2097
Participants | 50 | 52 |  | 48

9. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from first dose of study medication to 30 days after last dose of study medication (on-treatment), up to approximately 56 weeks.
  Deaths were collected in the post treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to approximately 10 years.
Time Frame: Pre-treatment deaths: Up to 14 days prior to treatment. On-treatment deaths: Up to 56 weeks. Post-treatment deaths: up to 10 years.
Population: Intent-to-Treat (ITT) Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab
Number analyzed (Participants) | 2093 | 2091 | 2100 | 2097
Participants
  Pre-treatment deaths | 1 | 2 | 1 | 2
  On-treatment deaths: number analyzed (Participants) | 2061 | 2076 | 2056 | 2076
  On-treatment deaths | 6 | 5 | 12 | 3
  Post-treatment deaths: number analyzed (Participants) | 2055 | 2071 | 2044 | 2073
  Post-treatment deaths | 189 | 190 | 250 | 228
  All deaths | 196 | 197 | 263 | 233

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 30 days post-treat follow-up, assessed up to approximately 56 weeks. Deaths were recorded from study start date until end of survival follow-up phase (end of study), assessed up to approximately 10 years.
Description: Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- Lapatinib Plus Trastuzumab: Lapatinib plus Trastuzumab: Events up to 30 days post-treatment
- Trastuzumab Followed by Lapatinib: Trastuzumab followed by Lapatinib: Events up to 30 days post-treatment
- Lapatinib: Lapatinib: Events up to 30 days post-treatment
- Trastuzumab: Trastuzumab: Events up to 30 days post-treatment
- Lapatinib Plus Trastuzumab (Post-Treatment): Lapatinib plus Trastuzumab (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
- Trastuzumab Followed by Lapatinib (Post-Treatment): Trastuzumab followed by Lapatinib (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
- Lapatinib (Post-Treatment): Lapatinib (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
- Trastuzumab (Post-Treatment): Trastuzumab (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
Arm/Group | Lapatinib Plus Trastuzumab | Trastuzumab Followed by Lapatinib | Lapatinib | Trastuzumab | Lapatinib Plus Trastuzumab (Post-Treatment) | Trastuzumab Followed by Lapatinib (Post-Treatment) | Lapatinib (Post-Treatment) | Trastuzumab (Post-Treatment)
All-Cause Mortality (participants affected / at risk) | 7/2093 | 7/2091 | 13/2100 | 5/2097 | 189/2055 | 190/2071 | 250/2044 | 228/2073
Serious Adverse Events (participants affected / at risk) | 379/2061 | 299/2076 | 394/2056 | 251/2076 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1930/2061 | 1862/2076 | 1887/2056 | 1649/2076 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Trastuzumab (N=2061) | Trastuzumab Followed by Lapatinib (N=2076) | Lapatinib (N=2056) | Trastuzumab (N=2076) | Lapatinib Plus Trastuzumab (Post-Treatment) (N=0) | Trastuzumab Followed by Lapatinib (Post-Treatment) (N=0) | Lapatinib (Post-Treatment) (N=0) | Trastuzumab (Post-Treatment) (N=0)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
ANAEMIA (Blood and lymphatic system disorders) | 7 | 6 | 13 | 7 | NA | NA | NA | NA
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 10 | 6 | 12 | 3 | NA | NA | NA | NA
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
LEUKOPENIA (Blood and lymphatic system disorders) | 20 | 4 | 13 | 7 | NA | NA | NA | NA
NEUTROPENIA (Blood and lymphatic system disorders) | 37 | 21 | 36 | 20 | NA | NA | NA | NA
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 1 | 2 | 7 | NA | NA | NA | NA
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
ATRIAL FIBRILLATION (Cardiac disorders) | 5 | 4 | 0 | 0 | NA | NA | NA | NA
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
ATRIAL THROMBOSIS (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
CARDIAC ARREST (Cardiac disorders) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 24 | 6 | 7 | 19 | NA | NA | NA | NA
CARDIAC VENTRICULAR THROMBOSIS (Cardiac disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
INTRACARDIAC THROMBUS (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 3 | 5 | 4 | 4 | NA | NA | NA | NA
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0 | 1 | 2 | NA | NA | NA | NA
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 | 0 | 0 | 1 | NA | NA | NA | NA
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PERICARDITIS (Cardiac disorders) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 1 | 0 | 0 | NA | NA | NA | NA
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
GILBERT'S SYNDROME (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
TINNITUS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
VERTIGO (Ear and labyrinth disorders) | 2 | 2 | 0 | 1 | NA | NA | NA | NA
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
GOITRE (Endocrine disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
HYPOTHYROIDISM (Endocrine disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
DIPLOPIA (Eye disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
PERIORBITAL OEDEMA (Eye disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
RETINAL DETACHMENT (Eye disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
ABDOMINAL MASS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 4 | 4 | 2 | NA | NA | NA | NA
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
COLITIS (Gastrointestinal disorders) | 4 | 0 | 1 | 1 | NA | NA | NA | NA
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | NA | NA | NA | NA
DIARRHOEA (Gastrointestinal disorders) | 53 | 6 | 44 | 9 | NA | NA | NA | NA
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ENTERITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
EPIPLOIC APPENDAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
GASTRITIS (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | NA | NA | NA | NA
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 1 | 0 | 4 | NA | NA | NA | NA
ILEUS (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | NA | NA | NA | NA
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | NA | NA | NA | NA
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
NAUSEA (Gastrointestinal disorders) | 5 | 3 | 7 | 6 | NA | NA | NA | NA
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
PANCREATITIS (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
REFLUX GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
VOLVULUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
VOMITING (Gastrointestinal disorders) | 9 | 3 | 9 | 8 | NA | NA | NA | NA
ADVERSE DRUG REACTION (General disorders) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
ASTHENIA (General disorders) | 2 | 0 | 4 | 1 | NA | NA | NA | NA
CHEST PAIN (General disorders) | 1 | 4 | 2 | 1 | NA | NA | NA | NA
CHILLS (General disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
CHRONIC FATIGUE SYNDROME (General disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
DEATH (General disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
DEVICE RELATED THROMBOSIS (General disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
FAT NECROSIS (General disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
FATIGUE (General disorders) | 5 | 2 | 7 | 2 | NA | NA | NA | NA
FEELING COLD (General disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
GRANULOMA (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
IMPAIRED HEALING (General disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
IMPLANT SITE THROMBOSIS (General disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
INFLAMMATION (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
LIPOGRANULOMA (General disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
MALAISE (General disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
MUCOSAL INFLAMMATION (General disorders) | 2 | 0 | 3 | 0 | NA | NA | NA | NA
NECROSIS (General disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
OEDEMA (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
OEDEMA PERIPHERAL (General disorders) | 0 | 2 | 0 | 1 | NA | NA | NA | NA
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PYREXIA (General disorders) | 11 | 16 | 13 | 5 | NA | NA | NA | NA
SUDDEN DEATH (General disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
BILIARY COLIC (Hepatobiliary disorders) | 0 | 2 | 0 | 1 | NA | NA | NA | NA
CHOLECYSTITIS (Hepatobiliary disorders) | 3 | 0 | 2 | 3 | NA | NA | NA | NA
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | NA | NA | NA | NA
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 2 | 0 | 0 | 1 | NA | NA | NA | NA
GALLBLADDER OBSTRUCTION (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 4 | 4 | 0 | NA | NA | NA | NA
HEPATIC LESION (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
HEPATITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HEPATOTOXICITY (Hepatobiliary disorders) | 3 | 3 | 5 | 0 | NA | NA | NA | NA
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 5 | 12 | 18 | 1 | NA | NA | NA | NA
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 74 | 55 | 86 | 11 | NA | NA | NA | NA
JAUNDICE (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | NA | NA | NA | NA
ANAPHYLACTIC REACTION (Immune system disorders) | 3 | 1 | 0 | 1 | NA | NA | NA | NA
ANAPHYLACTOID REACTION (Immune system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 2 | 0 | NA | NA | NA | NA
HYPERSENSITIVITY (Immune system disorders) | 4 | 4 | 1 | 4 | NA | NA | NA | NA
SARCOIDOSIS (Immune system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ACUTE HEPATITIS B (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
AMOEBIC DYSENTERY (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
ANAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
ANTIBIOTIC ASSOCIATED COLITIS (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ATYPICAL PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
BACTERAEMIA (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
BACTERIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
BREAST CELLULITIS (Infections and infestations) | 1 | 0 | 3 | 0 | NA | NA | NA | NA
BRONCHITIS (Infections and infestations) | 0 | 2 | 1 | 2 | NA | NA | NA | NA
BRONCHITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
CATHETER SITE CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
CELLULITIS (Infections and infestations) | 15 | 14 | 7 | 5 | NA | NA | NA | NA
CHEST WALL ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
CHLAMYDIAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
CONJUNCTIVITIS (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
CYSTITIS (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
DEVICE RELATED INFECTION (Infections and infestations) | 8 | 2 | 4 | 3 | NA | NA | NA | NA
DEVICE RELATED SEPSIS (Infections and infestations) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
DIVERTICULITIS (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
ERYSIPELAS (Infections and infestations) | 6 | 4 | 4 | 3 | NA | NA | NA | NA
GASTRIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
GASTROENTERITIS (Infections and infestations) | 3 | 3 | 3 | 1 | NA | NA | NA | NA
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
H1N1 INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HEPATITIS B (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
HEPATITIS C (Infections and infestations) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
HEPATITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
HERPES ZOSTER (Infections and infestations) | 1 | 2 | 3 | 0 | NA | NA | NA | NA
IMPLANT SITE CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
INFECTED CYST (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
INFECTED LYMPHOCELE (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
INFECTION (Infections and infestations) | 2 | 1 | 2 | 0 | NA | NA | NA | NA
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
LARGE INTESTINE INFECTION (Infections and infestations) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
LARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
LOCALISED INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 2 | 1 | 1 | NA | NA | NA | NA
LYMPH GLAND INFECTION (Infections and infestations) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
LYMPH NODE ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
LYMPHANGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
MALARIA (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
MASTITIS (Infections and infestations) | 2 | 1 | 6 | 2 | NA | NA | NA | NA
MENINGITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
NAIL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
NEUROBORRELIOSIS (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
OESOPHAGEAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
OSTEOMYELITIS (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
OVARIAN ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PARONYCHIA (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
PERITONITIS (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PNEUMOCYSTIS JIROVECII INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
PNEUMONIA (Infections and infestations) | 14 | 11 | 9 | 10 | NA | NA | NA | NA
PNEUMONIA ASPIRATION (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
PROGRESSIVE MULTIFOCAL LEUKOENCEPHALOPATHY (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
PYELONEPHRITIS (Infections and infestations) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 2 | 0 | NA | NA | NA | NA
SEPSIS (Infections and infestations) | 1 | 3 | 5 | 5 | NA | NA | NA | NA
SIALOADENITIS (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 2 | NA | NA | NA | NA
SKIN INFECTION (Infections and infestations) | 2 | 0 | 2 | 1 | NA | NA | NA | NA
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
STREPTOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 2 | 1 | 1 | NA | NA | NA | NA
SUPERINFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
TUBERCULOSIS (Infections and infestations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
TUBERCULOUS PLEURISY (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
URINARY TRACT INFECTION (Infections and infestations) | 2 | 6 | 2 | 7 | NA | NA | NA | NA
UROSEPSIS (Infections and infestations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
VIRAL INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
WOUND INFECTION (Infections and infestations) | 0 | 2 | 1 | 1 | NA | NA | NA | NA
WOUND INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | NA | NA | NA | NA
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
FOREIGN BODY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
FRACTURED COCCYX (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | NA | NA | NA | NA
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
RADIATION FIBROSIS - LUNG (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | NA | NA | NA | NA
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | NA | NA | NA | NA
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1 | NA | NA | NA | NA
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | NA | NA | NA | NA
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SEROMA (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1 | NA | NA | NA | NA
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | NA | NA | NA | NA
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
AMYLASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
BLOOD CREATININE INCREASED (Investigations) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
BLOOD MAGNESIUM DECREASED (Investigations) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
BLOOD UREA INCREASED (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
BLOOD URINE PRESENT (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
BODY TEMPERATURE INCREASED (Investigations) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
COAGULATION TEST ABNORMAL (Investigations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
EJECTION FRACTION DECREASED (Investigations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 4 | 3 | 0 | NA | NA | NA | NA
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
LIPASE (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
LIPASE INCREASED (Investigations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
LIVER FUNCTION TEST INCREASED (Investigations) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
PLATELET COUNT DECREASED (Investigations) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 0 | 3 | 0 | NA | NA | NA | NA
DEHYDRATION (Metabolism and nutrition disorders) | 11 | 3 | 12 | 4 | NA | NA | NA | NA
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | NA | NA | NA | NA
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HYPERPHOSPHATASAEMIA (Metabolism and nutrition disorders) | 4 | 4 | 1 | 0 | NA | NA | NA | NA
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | NA | NA | NA | NA
HYPOKALAEMIA (Metabolism and nutrition disorders) | 8 | 1 | 9 | 3 | NA | NA | NA | NA
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | NA | NA | NA | NA
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | NA | NA | NA | NA
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
CHEST WALL NECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
ACUTE PROMYELOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
BORDERLINE OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 3 | 4 | NA | NA | NA | NA
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2 | NA | NA | NA | NA
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
INTRADUCTAL PAPILLOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | NA | NA | NA | NA
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
LENTIGO MALIGNA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
OVARIAN GERM CELL TERATOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
SQUAMOUS CELL CARCINOMA OF THE VULVA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SUPERFICIAL SPREADING MELANOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2 | NA | NA | NA | NA
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
BRAIN HYPOXIA (Nervous system disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
CEREBELLAR ATAXIA (Nervous system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
DIZZINESS (Nervous system disorders) | 1 | 1 | 0 | 1 | NA | NA | NA | NA
EPILEPSY (Nervous system disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
FACIAL PARALYSIS (Nervous system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HEADACHE (Nervous system disorders) | 2 | 0 | 3 | 1 | NA | NA | NA | NA
HYPOTONIA (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
MIGRAINE (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
MOTOR NEURONE DISEASE (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 4 | 2 | 1 | NA | NA | NA | NA
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
POLYNEUROPATHY (Nervous system disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
QUADRIPARESIS (Nervous system disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
SEIZURE (Nervous system disorders) | 2 | 0 | 3 | 0 | NA | NA | NA | NA
SEROTONIN SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SYNCOPE (Nervous system disorders) | 2 | 1 | 3 | 5 | NA | NA | NA | NA
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
DEVICE DISLOCATION (Product Issues) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
DEVICE EXPULSION (Product Issues) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
THROMBOSIS IN DEVICE (Product Issues) | 1 | 1 | 1 | 0 | NA | NA | NA | NA
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
DEPRESSION (Psychiatric disorders) | 3 | 2 | 1 | 3 | NA | NA | NA | NA
INSOMNIA (Psychiatric disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
MENTAL DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SCHIZOPHRENIA (Psychiatric disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 1 | 1 | NA | NA | NA | NA
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
CALCULUS URINARY (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
NEPHRITIC SYNDROME (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 2 | 0 | 0 | NA | NA | NA | NA
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 2 | 1 | NA | NA | NA | NA
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ADENOMYOSIS (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
BREAST CALCIFICATIONS (Reproductive system and breast disorders) | 1 | 1 | 1 | 1 | NA | NA | NA | NA
BREAST DISORDER (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
BREAST FIBROSIS (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
BREAST HAEMATOMA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
BREAST INFLAMMATION (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
BREAST NECROSIS (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
BREAST SWELLING (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 4 | 1 | 3 | NA | NA | NA | NA
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 1 | 0 | 1 | NA | NA | NA | NA
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 6 | NA | NA | NA | NA
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | NA | NA | NA | NA
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | NA | NA | NA | NA
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | NA | NA | NA | NA
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | NA | NA | NA | NA
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 5 | NA | NA | NA | NA
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 2 | NA | NA | NA | NA
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ACNE (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | NA | NA | NA | NA
ANGIODERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | NA | NA | NA | NA
CUTANEOUS VASCULITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | NA | NA | NA | NA
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HYPERTROPHIC SCAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | NA | NA | NA | NA
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
RASH (Skin and subcutaneous tissue disorders) | 4 | 4 | 7 | 0 | NA | NA | NA | NA
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SKIN SWELLING (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | NA | NA | NA | NA
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 2 | 2 | 0 | NA | NA | NA | NA
EMBOLISM VENOUS (Vascular disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
FLUSHING (Vascular disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
HYPERTENSION (Vascular disorders) | 2 | 2 | 0 | 1 | NA | NA | NA | NA
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
HYPOTENSION (Vascular disorders) | 2 | 1 | 2 | 3 | NA | NA | NA | NA
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | NA | NA | NA | NA
RHEUMATOID VASCULITIS (Vascular disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 1 | NA | NA | NA | NA
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0 | NA | NA | NA | NA
THROMBOSIS (Vascular disorders) | 2 | 2 | 1 | 2 | NA | NA | NA | NA
VASCULAR INSUFFICIENCY (Vascular disorders) | 1 | 0 | 0 | 0 | NA | NA | NA | NA
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 1 | 0 | 0 | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Trastuzumab (N=2061) | Trastuzumab Followed by Lapatinib (N=2076) | Lapatinib (N=2056) | Trastuzumab (N=2076) | Lapatinib Plus Trastuzumab (Post-Treatment) (N=0) | Trastuzumab Followed by Lapatinib (Post-Treatment) (N=0) | Lapatinib (Post-Treatment) (N=0) | Trastuzumab (Post-Treatment) (N=0)
ANAEMIA (Blood and lymphatic system disorders) | 226 | 168 | 169 | 223 | NA | NA | NA | NA
LEUKOPENIA (Blood and lymphatic system disorders) | 174 | 138 | 155 | 168 | NA | NA | NA | NA
NEUTROPENIA (Blood and lymphatic system disorders) | 233 | 175 | 220 | 179 | NA | NA | NA | NA
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 59 | 46 | 45 | 107 | NA | NA | NA | NA
ABDOMINAL PAIN (Gastrointestinal disorders) | 146 | 108 | 148 | 79 | NA | NA | NA | NA
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 137 | 111 | 110 | 78 | NA | NA | NA | NA
CONSTIPATION (Gastrointestinal disorders) | 120 | 184 | 135 | 156 | NA | NA | NA | NA
DIARRHOEA (Gastrointestinal disorders) | 1516 | 1039 | 1278 | 399 | NA | NA | NA | NA
DYSPEPSIA (Gastrointestinal disorders) | 174 | 140 | 156 | 116 | NA | NA | NA | NA
NAUSEA (Gastrointestinal disorders) | 393 | 393 | 381 | 285 | NA | NA | NA | NA
STOMATITIS (Gastrointestinal disorders) | 203 | 141 | 161 | 98 | NA | NA | NA | NA
VOMITING (Gastrointestinal disorders) | 251 | 181 | 215 | 151 | NA | NA | NA | NA
ASTHENIA (General disorders) | 202 | 178 | 175 | 171 | NA | NA | NA | NA
FATIGUE (General disorders) | 511 | 515 | 443 | 439 | NA | NA | NA | NA
MUCOSAL INFLAMMATION (General disorders) | 227 | 149 | 164 | 114 | NA | NA | NA | NA
OEDEMA PERIPHERAL (General disorders) | 144 | 149 | 138 | 160 | NA | NA | NA | NA
PYREXIA (General disorders) | 227 | 188 | 132 | 171 | NA | NA | NA | NA
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 96 | 103 | 121 | 31 | NA | NA | NA | NA
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 348 | 378 | 366 | 281 | NA | NA | NA | NA
NASOPHARYNGITIS (Infections and infestations) | 128 | 111 | 96 | 150 | NA | NA | NA | NA
PARONYCHIA (Infections and infestations) | 262 | 165 | 206 | 22 | NA | NA | NA | NA
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 117 | 96 | 93 | 118 | NA | NA | NA | NA
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 91 | 127 | 82 | 129 | NA | NA | NA | NA
DECREASED APPETITE (Metabolism and nutrition disorders) | 223 | 173 | 188 | 142 | NA | NA | NA | NA
HYPERPHOSPHATASAEMIA (Metabolism and nutrition disorders) | 81 | 109 | 120 | 76 | NA | NA | NA | NA
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 340 | 348 | 320 | 451 | NA | NA | NA | NA
BACK PAIN (Musculoskeletal and connective tissue disorders) | 128 | 133 | 119 | 126 | NA | NA | NA | NA
BONE PAIN (Musculoskeletal and connective tissue disorders) | 87 | 109 | 91 | 122 | NA | NA | NA | NA
MYALGIA (Musculoskeletal and connective tissue disorders) | 211 | 214 | 174 | 252 | NA | NA | NA | NA
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 135 | 125 | 98 | 175 | NA | NA | NA | NA
DIZZINESS (Nervous system disorders) | 104 | 127 | 115 | 118 | NA | NA | NA | NA
HEADACHE (Nervous system disorders) | 192 | 241 | 161 | 262 | NA | NA | NA | NA
NEUROPATHY PERIPHERAL (Nervous system disorders) | 177 | 183 | 173 | 178 | NA | NA | NA | NA
PARAESTHESIA (Nervous system disorders) | 125 | 110 | 107 | 131 | NA | NA | NA | NA
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 164 | 159 | 162 | 194 | NA | NA | NA | NA
INSOMNIA (Psychiatric disorders) | 168 | 172 | 152 | 190 | NA | NA | NA | NA
COUGH (Respiratory, thoracic and mediastinal disorders) | 219 | 201 | 153 | 242 | NA | NA | NA | NA
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 147 | 146 | 103 | 170 | NA | NA | NA | NA
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 319 | 213 | 244 | 165 | NA | NA | NA | NA
ACNE (Skin and subcutaneous tissue disorders) | 134 | 138 | 112 | 20 | NA | NA | NA | NA
ALOPECIA (Skin and subcutaneous tissue disorders) | 109 | 135 | 110 | 151 | NA | NA | NA | NA
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 117 | 96 | 124 | 19 | NA | NA | NA | NA
DRY SKIN (Skin and subcutaneous tissue disorders) | 262 | 244 | 280 | 86 | NA | NA | NA | NA
ERYTHEMA (Skin and subcutaneous tissue disorders) | 122 | 104 | 93 | 87 | NA | NA | NA | NA
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 359 | 272 | 294 | 220 | NA | NA | NA | NA
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 181 | 105 | 126 | 47 | NA | NA | NA | NA
PRURITUS (Skin and subcutaneous tissue disorders) | 316 | 268 | 334 | 134 | NA | NA | NA | NA
RASH (Skin and subcutaneous tissue disorders) | 771 | 685 | 767 | 223 | NA | NA | NA | NA
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 145 | 98 | 123 | 7 | NA | NA | NA | NA
HOT FLUSH (Vascular disorders) | 211 | 225 | 190 | 272 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.